CLINICAL TRIAL: NCT01607658
Title: A Placebo-Controlled, Randomized, Double-Blind, Parallel-Group, Dose-Finding Trial to Evaluate the Efficacy and Safety of TBS-2 Intranasal Testosterone Gel in Women With Acquired Female Orgasmic Disorder
Brief Title: Efficacy and Safety of TBS-2 Testosterone Gel in Women With Acquired Female Orgasmic Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Acerus Pharmaceuticals Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TBS-2-AMB-2012-01
Record Dates: First submitted 2012-05-18; First posted 2012-05-30 (Estimated); Results first posted 2018-08-13 (Actual); Last update posted 2018-08-13 (Actual); Status verified 2018-08

CONDITIONS: Female Orgasmic Disorder
Keywords: Testosterone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Placebo (Placebo Comparator): Placebo intranasal gel administered prn, 2-8 hours before a planned sexual event
  Interventions: Drug: Placebo
- Experimental 1 (Experimental): Low dose TBS-2 (0.6 mg) testosterone intranasal gel administered prn
  Interventions: Drug: Low dose TBS-2
- Experimental 2 (Experimental): Medium dose TBS-2 (1.2 mg) testosterone intranasal gel administered prn
  Interventions: Drug: Medium dose TBS-2
- Experimental 3 (Experimental): High dose TBS-2 (1.8 mg) testosterone intranasal gel administered prn
  Interventions: Drug: High dose TBS-2

INTERVENTIONS:
Drug: Placebo — placebo intranasal gel administered prn, 2-8 hours before a planned sexual event
  Arms: Placebo
Drug: Low dose TBS-2 — Low dose testosterone intranasal gel administered prn 2-8 hrs before a planned sexual event
  Arms: Experimental 1
Drug: Medium dose TBS-2 — Medium dose testosterone intranasal gel administered prn 2-8 hrs before a planned sexual event
  Arms: Experimental 2
Drug: High dose TBS-2 — High dose testosterone intranasal gel administered prn 2-8 hrs before a planned sexual event
  Arms: Experimental 3

SUMMARY:
The purpose of this study is to assess and compare the effects of 3 dose strengths of TBS-2 intranasal testosterone gel to placebo on the occurrence of orgasm.

ELIGIBILITY:
Inclusion Criteria

Subjects who meet the following criteria may be included in the study:

At Visit 1:≤

* Be a generally healthy female aged 18 years and older, inclusive, who has no physical impediment to sexual function
* Have a diagnosis of acquired female orgasmic disorder defined as absence of orgasm during the past 6 months and according to the Diagnostic and Statistical Manual of Mental Disorders IV (DSM-IV) criteria. Subtype should be generalized and not due to etiological factors that would be unlikely to be related to hormone function (eg, depression, relationship discord, alcoholism, surgery, injury). Hypoactive sexual desire disorder as a co-morbid disorder is allowed only if it began after the female orgasmic disorder diagnosis;
* Have a score of >15 with a score of ≥2 for question #15 on the FSDS DAO at Screening Visit;
* Be a sexually active, hetero- or homosexual woman in a steady relationship for at least 6 months and agree to have at least 4 sexual events over 28-day period of time. The subject's partner should not have any untreated sexual dysfunctions;
* Be on a reliable birth control method (ie, stable systemic hormonal contraception for the whole duration of the study and 30 days after study completion [for at least 3 months prior to study], IUD, barrier method) or not engaging in heterosexual intercourse. Birth control method used by subject at screening is not to be changed during the course of the study;
* Have a normal ENT examination;
* Have a body mass index ≤35;
* Have a clinically acceptable pelvic examination and Pap smear as read by a licensed laboratory facility (no evidence of malignancy) within the 2 years prior to Randomization;
* Have a clinically acceptable mammogram;
* Be able to complete a web-based questionnaire within 24 hours of each sexual event;
* Be able to read English and provide written informed consent; and

At Visit 2:

* Have at least 4 sexual events and an absence of orgasm during the 28 day Screening/Baseline Period as determined by MONASH WHP FSSQ.

Exclusion Criteria

Subjects who meet any of the following criteria will not be eligible to participate in the study:

* Have a known history of hypersensitivity to testosterone or any component of the study drug;
* Have a history of any clinically relevant psychiatric disorder that could impact sexual functioning, contribute to increased risk for patient safety, or significantly compromise participation in the study (eg, bipolar disorders, psychotic disorders, severe anxiety, eating disorders, borderline personality disorder, untreated Major Depressive Disorder);
* Have a score of ≥14 on the Beck Depression Inventory II at Screening Visit. Subjects with a score of ≥14 and ≤19 at Screening may be eligible to participate in the study if a specialist (psychologist or psychiatrist) concludes that the subject is not clinically depressed;
* Have other concurrent female sexual dysfunction disorders as defined by DSM-IV criteria, eg, Sexual Aversion Disorder, Substance-Induced sexual dysfunction, dyspareunia (not caused by inadequate foreplay stimulation or alleviated by lubricants), vaginismus, Gender Identity Disorder, paraphilia, or sexual dysfunction due to a general medical condition;
* Be experiencing relational discord;
* Have a history of dementia or other neurodegenerative diseases, organic brain disease, stroke, transient ischemic attacks, brain surgery, significant brain trauma, multiple sclerosis, spinal cord injury, peripheral neuropathy, and epilepsy (febrile seizures limited to childhood do not exclude patients);
* Be currently receiving treatment with selective norepinephrine reuptake inhibitors (SNRIs) and selective serotonin reuptake inhibitors (SSRIs) and/or medications that interfere with the metabolism of testosterone (eg, anastrozole, clomiphene, testolactone, ketoconazole, spironolactone, histamine 2 [H2 receptor blockers, etc.]);
* Have a history of, or current evidence of, abuse of alcohol or any drug substance, licit or illicit, or be a regular drinker of more than 3 units of alcohol daily (1 unit = 300 mL beer, 1 glass wine, 1 measure spirit);
* Have a history of cancer other than nonmelanotic skin cancer;
* Have a history of deep venous thrombosis or coagulation disorders;
* Have a significant medical condition (eg, hepatic, renal cardiovascular, endocrine including diabetes mellitus). Subjects with treated hypertension, treated hyperlipidemia, or treated thyroid disease will not be excluded provided they have been on stable therapy for at least 3 months;
* Had any major surgical procedure within the past 6 months including hysterectomy, hysterectomy with bilateral salpingo oophorectomy, or vaginal incontinence surgery
* Are receiving treatment with systemic glucocorticosteroids, sex steroid hormones such as androgens (eg, dehydroepiandrosterone [DHEA]) or gestagens (eg, anabolic steroids) and using any post menopausal hormone therapy;
* Have a history of severe or multiple drug allergies, severe adverse drug reaction or drug-related leucopenia;
* Have a history of nasal disorders (eg, atrophic rhinitis, polyposis, abuse of nasal decongestants, clinically relevant nasal septum deviation, recurrent epistaxis), sinus disease or nasal surgery and/or seasonal or perennial allergic rhinitis in the active phase;
* Be using any form of chronic intranasal medication delivery, specifically nasal corticosteroids or decongestants;
* Have a diagnosis of sleep apnea and be using a continuous positive airway pressure/automatic positive airway device;
* Have a history of diagnosed hirsutism, alopecia or clinically significant acne;
* Have a history of diagnosed polycystic ovarian syndrome;
* Have pelvic inflammatory disease, chronic urinary tract, vaginal, or cervical infections, interstitial cystitis, vulvodynia, or significant symptomatic vaginal atrophy;
* Are currently pregnant, by history or positive serum pregnancy test at Screening Visit or have been pregnant within the 12 months prior to Screening Visit;
* Is breast feeding or have breast fed within the 6 months prior to Screening Visit;
* Are positive for hepatitis B-surface antigen, hepatitis C, or Human Immunodeficiency Virus (HIV);
* Have abnormal thyroid stimulating hormone level;
* For pre-menopausal women, have SHBG value <18 86 nmol/L; For post-menopausal women, have SHBG value >160 nmol/L
* Have any medical or psychiatric condition, physical examination finding, or laboratory result which, in the opinion of the principal investigator, would put the subject at additional medical risk or make her unlikely to be able to comply with study requirements; or
* Have received any drug as part of a research study within 30 days prior to the Screening Visit.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 253 (Actual)
Dates: Start 2012-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Natalia Tkachenko, MD, Study Director — Trimel Pharmaceuticals Corporation
Locations (53):
- United States (43):
  - Radiant Research, Birmingham, Alabama
  - Medical Affiliated Research Center Inc., Huntsville, Alabama
  - Radiant Research Inc., Chandler, Arizona
  - Quality of Life Medical Research Center, Tucson, Arizona
  - Medical Center for Clinical Research, San Diego, California
  - San Diego Sexual Medicine, San Diego, California
  - Downtown Women's Health Care, Denver, Colorado
  - Radiant Research Inc., Denver, Colorado
  - Thameside OB/GYN Centre, Groton, Connecticut
  - Greater Hartford Women's Health Associates, Hartford, Connecticut
  - Tampa Bay Medical Research Inc., Clearwater, Florida
  - Clinical Research of South Florida, Coral Gables, Florida
  - Clinical Physiology Associates, Fort Myers, Florida
  - University of Florida - Jacksonville, Jacksonville, Florida
  - Compass Research East LLC, Oviedo, Florida
  - Center for Marital and Sexual Health of South Florida, West Palm Beach, Florida
  - Atlanta North Gynecology, PC, Roswell, Georgia
  - Women's Health Practice, Champaign, Illinois
  - Radiant Research Inc., Chicago, Illinois
  - Radiant Reseach, Overland Park, Kansas
  - Maryland Center for Sexual Health, Lutherville, Maryland
  - QUEST Research Institute, Bingham Farms, Michigan
  - Radiant Research Inc., Edina, Minnesota
  - Montana Health Research Institute, Billings, Montana
  - Womens Clinic of Lincoln P.C., Lincoln, Nebraska
  - Columbia University School of Nursing, New York, New York
  - Wake Research Associates LLC, Raleigh, North Carolina
  - Lillestol Research LLC, Fargo, North Dakota
  - Radiant Research, Akron, Ohio
  - Center for Marital and Sexual Health Inc., Beachwood, Ohio
  - Columbus Center for Women's Health Research, Columbus, Ohio
  - University Hospitals Case Medical Center, Mayfield Heights, Ohio
  - Cincinnati Urogynecology Associates (TRIHEALTH), West Chester, Ohio
  - Clinical Research of Philadelphia LLC, Philadelphia, Pennsylvania
  - Clinical Research Associates, Inc, Nashville, Tennessee
  - Radiant Research Inc., Dallas, Texas
  - Texas Diabetes and Endocrinology, Round Rock, Texas
  - Radiant Research Inc., San Antonio, Texas
  - San Antonio Psychiatric Research Center Dba Croft Group Research Center, San Antonio, Texas
  - University of Virginia Center for Psychiatric Clinical Research, Charlottesville, Virginia
  - Virginia Research Center, Midlothian, Virginia
  - Tidewater Physicians for Women, Norfolk, Virginia
  - Women's Clincial Research Center, Seattle, Washington
- Australia (4):
  - Monash University, Melbourne
  - Keogh Institute for Medical Research, Nedlands
  - The Robinson Institute University of Adelaide, North Adelaide
  - Barbara Gross Research Unit, Randwick
- Canada (6):
  - Alta Clinical Research Inc., Edmonton, Alberta
  - Gain Medical Centre, Coquitlam, British Columbia
  - Discovery Clinical Services, Ltd, Victoria, British Columbia
  - Victoria Clinical Research Inc, Victoria, British Columbia
  - Manitoba Clinic, Winnipeg, Manitoba
  - Manna Research, Toronto, Ontario

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Dose TBS-2: Low dose TBS-2 (0.6 mg) testosterone intranasal gel administered prn
  Low dose TBS-2: Low dose testosterone intranasal gel administered prn 2-8 hrs before a planned sexual event
- Medium Dose TBS-2: Medium dose TBS-2 (1.2 mg) testosterone intranasal gel administered prn
  Medium dose TBS-2: Medium dose testosterone intranasal gel administered prn 2-8 hrs before a planned sexual event
- High Dose TBS-2: High dose TBS-2 (1.8 mg) testosterone intranasal gel administered prn
  High dose TBS-2: High dose testosterone intranasal gel administered prn 2-8 hrs before a planned sexual event
Period: Overall Study
Arm/Group | Placebo | Low Dose TBS-2 | Medium Dose TBS-2 | High Dose TBS-2
Started | 65 | 67 | 58 | 63
Completed | 56 | 56 | 47 | 52
Not Completed | 9 | 11 | 11 | 11

BASELINE CHARACTERISTICS:
Population: ITT population
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Low Dose TBS-2 | Medium Dose TBS-2 | High Dose TBS-2 | Total
Number analyzed (Participants) | 65 | 67 | 58 | 63 | 253
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.4 (12.36) | 44.5 (12.09) | 44.3 (11.64) | 42.4 (11.47) | 43.4 (11.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 65 | 67 | 58 | 63 | 253
  Male | 0 | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 10 | 6 | 9 | 28
  Not Hispanic or Latino | 62 | 57 | 52 | 54 | 225
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 2 | 0 | 1 | 3
  Asian | 2 | 0 | 0 | 3 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 14 | 11 | 11 | 10 | 46
  White | 47 | 51 | 46 | 47 | 191
  More than one race | 2 | 2 | 1 | 1 | 6
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 3 | 3 | 4 | 4 | 14
  United States | 53 | 58 | 48 | 55 | 214
  Australia | 9 | 6 | 6 | 4 | 25

OUTCOME MEASURES:

1. Primary Outcome: Number of Orgasms Over an 84 Day Period Compared to Placebo Over the Entire Treatment Period
Time Frame: 84 days
Population: ITT Population
Measure: Mean (Standard Deviation); unit: orgasms
Arm/Group | Placebo | Low Dose TBS-2 | Medium Dose TBS-2 | High Dose TBS-2
Number analyzed (Participants) | 65 | 67 | 58 | 63
orgasms | 2.8 (4.60) | 3.9 (5.22) | 3.2 (4.70) | 1.9 (3.47)

2. Secondary Outcome: Change in Sexual Event Satisfaction Over a 28-day Period (Day 57 to Day 84) Compared to Baseline (Day -28 to Day 0)
Description: as measured by Monash Women's Health Program Female Sexual Satisfaction Questionnaire (MONASH WHP FSSQ) question 11.
  MONASH WHP FSSQ question 11 asks participants to comment on how satisfying they found the sex to be from "Not at all" to "Very much so". The lowest score is 1 and the highest is 9. All scores for each 28-day period were averaged. Change from baseline was obtained by subtracting baseline 28-day average from the 28-day period at the end of the study (Day 57 to 84).
Time Frame: Baseline (Day -28 to Day 0) and End of Study (Day 57 to 84)
Population: The number of participants analyzed is equal to the number of participants who completed the Day 84 visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Low Dose TBS-2 | Medium Dose TBS-2 | High Dose TBS-2
Number analyzed (Participants) | 54 | 55 | 47 | 54
units on a scale | 1.37 (1.624) | 1.52 (1.586) | 1.59 (1.803) | 1.27 (1.707)

3. Secondary Outcome: Change in Distress Due to Female Orgasmic Disorder From Day 0 Baseline to Day 84
Description: as measured by Female Sexual Distress Scale (FSDS-DAO) Question #15 on Day 0 and 84, respectively. Question #15 evaluates the level of distress related to problems with orgasm. It is rated on a 5-point Likert scale (from 0 to 4, i.e. never [0], rarely [1], occasionally [2], frequently [3], or always [4]). Higher scores indicate more distress.
Time Frame: Day 0 and Day 84
Population: The number of participants analyzed is equal to the number of participants who completed the Day 84 visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Low Dose TBS-2 | Medium Dose TBS-2 | High Dose TBS-2
Number analyzed (Participants) | 56 | 56 | 47 | 53
units on a scale | -0.9 (1.09) | -1.3 (1.40) | -0.9 (1.10) | -0.8 (1.23)

4. Secondary Outcome: Change in Global Sexual Functioning From Day 0 to Day 84
Description: as measured by Female Sexual Function Index (FSFI) on Day 0 and 84, respectively. The FSFI, a 19-item questionnaire, has been developed as a brief, multidimensional self-report instrument for assessing the key dimensions of sexual frustration in women. The questionnaire provides scores on 6 domains of sexual function (desire, arousal, lubrication, orgasm, satisfaction, and pain) as well as a total score. Fifteen items are rated on a 6-point Likert scale (from 0 to 5) and 4 items on a 5-point Likert scale (from 1 to 5). The scores are added and converted using a conversion factor so that the maximum score for each domain is 6. The overall FSFI score can range from 2 to 36. Higher scores indicate better or higher sexual function.
Time Frame: Day 0 and Day 84
Population: The number of participants analyzed is equal to the number of participants who completed the Day 84 visit.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Low Dose TBS-2 | Medium Dose TBS-2 | High Dose TBS-2
Number analyzed (Participants) | 53 | 55 | 47 | 54
units on a scale | 2.90 (5.622) | 3.42 (6.278) | 3.33 (6.707) | 3.35 (5.835)

ADVERSE EVENTS:
Time Frame: 84 days
Arm/Group | Placebo | Low Dose TBS-2 | Medium Dose TBS-2 | High Dose TBS-2
All-Cause Mortality (participants affected / at risk) | 0/65 | 0/67 | 0/58 | 0/63
Serious Adverse Events (participants affected / at risk) | 0/65 | 0/67 | 0/58 | 0/63
Other Adverse Events (participants affected / at risk) | 24/65 | 35/67 | 20/58 | 38/63
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=65) | Low Dose TBS-2 (N=67) | Medium Dose TBS-2 (N=58) | High Dose TBS-2 (N=63)
Upper Respiratory Tract Infection (Infections and infestations) | 4 | 5 | 2 | 7
Nasopharyngitis (Infections and infestations) | 5 | 0 | 1 | 0
Urinary Tract Infection (Infections and infestations) | 2 | 0 | 3 | 1
Pharyngitis (Infections and infestations) | 1 | 2 | 0 | 1
Sinusitis (Infections and infestations) | 3 | 0 | 0 | 1
Nasal Inflamation (Respiratory, thoracic and mediastinal disorders) | 2 | 4 | 2 | 5
Nasal Discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 5
Nasal Mucosal Disorder (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 1 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 1 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 4 | 3 | 5
Hair Growth Abnormal (Skin and subcutaneous tissue disorders) | 1 | 3 | 0 | 5
Hirsutism (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 3
Scab (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 3
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 0
Urine Analysis Abnormal (Investigations) | 0 | 0 | 2 | 0
Contusion (Injury, poisoning and procedural complications) | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 1 | 2 | 0 | 2
Fatigue (General disorders) | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes